CLINICAL TRIAL: NCT06002347
Title: Development, Acceptability, and Short-Term Outcomes of a Parent Module for a Brief, Bullying Bystander Intervention for Middle School Students in Rural, Low-Income Communities
Brief Title: Middle School Parent Module for a Brief Bullying Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boise State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Aida Midgett, Professor, Boise State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 101-SB21-051; 5U54GM104944 (NIH)
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Bullying
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STAC Parent Module (Experimental)
  Interventions: Behavioral: STAC Parent Module for Middle School

INTERVENTIONS:
Behavioral: STAC Parent Module for Middle School — The STAC Parent Module is a 30-minute pre-recorded online presentation that includes normative feedback, didactic information, a review of the student STAC strategies and corresponding strategies parents can use to support students who act as defenders, and information about "perceptions vs. facts" about bullying.

SUMMARY:
This study evaluates the feasibility and short-term outcomes of a parent training designed as a companion module to a bullying bystander intervention (STAC) for middle school students in rural communities. The aim of this project is to provide a brief, low-cost intervention that can be easily disseminated as part of a school-based bullying prevention program to address this important public health problem.

ELIGIBILITY:
Inclusion Criteria:

1. Being a parent of an adolescent enrolled in grades 6, 7, or 8 in a participating middle school in Idaho.
2. Speaks and reads English.
3. Consents to participate.

Exclusion Criteria:

1. Speaks and reads only a language other than English.
2. Does not consent for participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boise State Univerity, Boise, Idaho, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STAC Parent Module
Started | 23
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.17 (7.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Knowledge and Confidence to Support Defenders
Description: Modified version of Teacher-Advocates Pre- and Post-Scale (TAPPS) Knowledge and confidence to support defenders was measured using a modified version of the TAPPS. The TAPPS is an 11 item survey that measures knowledge of buying behaviors, knowledge of how to support students using the STAC strategies, and confidence supporting students who intervene in bullying situations. Items are rated on a 4-point Likert Scale ranging from 1 (Totally Disagree) to 4 (Totally Agree) and were summed to compute a total scale score.
  Minimum =11; Maximum = 44
  Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
score on a scale
  Pre-Test | 33.52 (3.90)
  Post-Test | 38.90 (4.36)

2. Primary Outcome: Confidence Managing Bullying
Description: Modified version of Teacher's Attitudes about Bullying Questionnaire Confidence about managing bullying was measured using a modified version of the Teacher's Attitudes about Bullying Questionnaire. This questionnaire is a 22 item survey. The 3-item Confidence in Managing Bullying Subscale was used. Items are rated on a 5-point Likert Scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree) and are summed to compute a total scale score.
  Minimum = 3; Maximum = 15
  Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
score on a scale
  pre-test | 12.00 (2.00)
  post-test | 13.75 (1.21)

3. Primary Outcome: Comfort Managing Bullying
Description: National Education Association Bullying Survey Parent comfort with managing bullying was measured using items from the National Education Association Bullying Survey. Parents were asked "How comfortable would the participant feel intervening when the participant sees the following bullying behaviors?" followed by five types of bullying (a) Physical, (b) Verbal, (c) Relational, (d) Cyberbullying, and (e) Sexting . Items are rated on a 5-point Likert Scale ranging from 1 (Very Uncomfortable) to 5 (Very Comfortable) and are summed to compute a total scale score.
  Minimum = 5; Maximum = 25
  Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
score on a scale
  pre-test | 11.04 (3.67)
  post-test | 13.70 (1.84)

4. Primary Outcome: Parental Role
Description: National Education Association Bullying Survey Parental role in handling bullying situations was measured by four items from the National Education Association Bullying Survey. Items are rated on a 4-point Likert Scale ranging from 1 (Strongly Disagree) to 4 (Strongly Agree) and are summed to create the scale.
  Minimum = 4; Maximum = 16
  Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
score on a scale
  pre-test | 12.17 (2.27)
  post-test | 13.95 (2.09)

5. Primary Outcome: Bullying Self-Efficacy
Description: Bullying Self-Efficacy Parents' perceptions of ability to help the participants' child respond to bullying were measured using a 6-item scale. Items are rated on a 4-point Likert Scale ranging from 1 (Not at All) to 4 (A Lot) and are summed to create the scale.
  Minimum = 6; Maximum = 24
  Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
score on a scale
  pre-test | 20.44 (2.37)
  post-test | 22.50 (1.67)

6. Primary Outcome: Communication Self-Efficacy
Description: Communication Self-Efficacy Parents' self-efficacy to talk with the participants' child about bullying was assessed using a 6-item scale. Items are rated on a 5-point Likert Scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree) and are summed to create the scale.
  Minimum = 6; Maximum = 30
  Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
score on a scale
  pre-test | 25.39 (3.01)
  post-test | 27.75 (2.27)

7. Primary Outcome: Attitudes About Bullying
Description: Provictim Scale Attitudes about bullying were measured using the Provictim Scale, including 6 items that reflect anti-bullying attitudes. Items are rated on a 5-point Likert Scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree) and are summed to create the scale.
  Minimum = 6; Maximum = 30
  Higher scores are better outcomes
Time Frame: pre-training (baseline); immediate post-training (30 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
score on a scale
  pre-test | 24.22 (2.81)
  post-test | 25.65 (3.12)

8. Primary Outcome: Intention to Use Parent STAC Strategies
Description: Use of STAC Strategies The intention to use Parent STAC strategies was measured using an adapted version of the Use of STAC Strategies for students and teachers. The 4-item measure asks parents "How likely is the participant to use these strategies to support the participants' adolescent to intervene in bullying in the future? a) Stealing the Show - support adolescents to use humor or distraction to get the attention away from the bullying situation, b) Turning it Over - support adolescents who tell the participant about bullying or support adolescents to report to an adult at school, c) Accompanying Others - support adolescents who reach out to a student who was a target of bullying, and d) Coaching Compassion - support adolescents who help the student who bullied develop empathy for the target." Items are rated on a 5-point Likert Scale ranging from 1 (Very Unlikely) to 5 (Very Likely).
Time Frame: immediate post-training (30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
Participants
  Stealing the Show | 14
  Turning it Over | 19
  Accompanying Others | 19
  Coaching Compassion | 19

9. Secondary Outcome: Acceptability of the Parent STAC Training
Description: Acceptability of the Parent STAC Training Program acceptability (e.g., how easy the program is to understand, utility of the program, program characteristics including interesting content and relevance of information and examples presented, participant learning, and interest in recommending program to others) was assessed using a social validity survey composed of 7 items. Items were ranked on a 4-point scale from 1 (Strongly Disagree) to 4 (Strongly Agree).
Time Frame: immediate post-training (30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
Participants
  Easy to understand | 20
  Useful | 18
  Interesting | 18
  Information Relevant | 19
  Examples Relevant | 20
  Learned something | 18
  Would recommend | 19

10. Secondary Outcome: Interest in Receiving Bullying Prevention
Description: Interest in Receiving Bullying Prevention Participants were asked the question "how interested the participant would be in receiving a bullying prevention program." Responses were rated on a 5-point response scale with anchors ranging from 1 (Not at all Interested) to 5 (Extremely Interested).
Time Frame: immediate post-training (30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
Participants | 20

11. Secondary Outcome: Features of a Technology-Based Program
Description: Features of A Technology-Based Program Participants were asked a series of questions regarding features (e.g., interactive, self-paced, based on research, designed by a reputable institution, containing slides, fact sheets, and quizzes) of a technology-based program. Items were rated on a 5-point scale from 1 (Not at All Important) to 5 (Extremely Important). The criteria for a participant to be counted as perceiving the feature to be important was for the participant to select the response rating 3 (Important), 4 (Very Important), or 5 (Extremely Important).
Time Frame: immediate post-training (30 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | STAC Parent Module
Number analyzed (Participants) | 20
Participants
  Interactive | 14
  Self-paced | 18
  Based on research | 20
  Designed by reputable institution | 18
  Have slides, fact sheets, and graphics | 15
  Have quizzes | 10

ADVERSE EVENTS:
Time Frame: 12 days
Arm/Group | STAC Parent Module
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT06002347/Prot_SAP_000.pdf